CLINICAL TRIAL: NCT00628108
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Parallel-Group Study of the Safety of Levocetirizine Dihydrochloride Oral Liquid Formulation in Children Aged 6 Months to 11 Months With Symptoms of Allergic Rhinitis or Chronic Urticaria.
Brief Title: Safety Study of Levocetirizine Dihydrochloride Oral Liquid Formulation in Children Aged 6 Months to 11 Months
Acronym: BALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A00423; RPCE08K2403; 2007-003458-28 (EudraCT Number)
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Rhinitis; Chronic Urticaria
Keywords: Xyzal; Levocetirizine; Allergy; Children; Seasonal Allergies
MeSH Terms: conditions — Rhinitis, Allergic; Chronic Urticaria; Hypersensitivity; Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Levocetirizine (Experimental)
  Interventions: Drug: Levocetirizine 1.25 mg

INTERVENTIONS:
Drug: Levocetirizine 1.25 mg — Levocetirizine dihydrochloride 1.25 mg (5 drops containing 5 mg/mL) dosed once a day for 2 weeks
  Other Names: Xyzal
  Arms: Levocetirizine
Other: Placebo — Placebo oral liquid once a day for two weeks
  Arms: Placebo

SUMMARY:
To determine the safety of levocetirizine in children ages 6-11 months with symptoms of allergic rhinitis or chronic idiopathic urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, male or female pediatric subject, aged from 6 to 11 months (6 months - < 1 year) at the randomization visit
* The subject must present at least one symptom most commonly associated with allergic rhinitis or chronic idiopathic urticaria
* Candidate for antihistamine treatment or received antihistamine in the past for similar symptoms as those presenting

Exclusion Criteria:

* Any clinically significant medical condition or abnormality other than the primary diagnosis for which an antihistamine is indicated
* Be initiating or changing the dose of an immunotherapy regimen during the course of the study (Visit 1 to Visit 4)
* Any Electrocardiogram (ECG) parameters, including a QTcF interval > 443 msec measured by an ECG obtained at the Screening Visit, outside the normal reference ranges
* Any clinical laboratory tests performed at Screening Visit, other than those related with the allergic condition, outside the reference ranges. Subjects having values outside the accepted reference range can be included if in the Investigator's opinion, they are of no clinical significance
* Personal history of seizure, febrile seizure or sleep apnea
* Below the lower 5th or above 95th percentile for body weight and/or height based upon CDC Growth Charts for Body Weight and Length
* Allergy or intolerance to levocetirizine dihydrochloride or its excipients, or to any other piperazine derivatives, such as hydroxyzine, cetirizine, cyclizine, meclozine, buclizine
* Current or past intake (including exposure through breast milk) of the following medications within the specified wash-out period before the Randomization Visit (V2):

  * Systemic corticosteroids within the past 28 days
  * Leukotriene-receptor antagonists (e.g. montelukast [Singulair] or zafirlukast [Accolate] within the past 7 days)
  * Mast-cell stabilizers (e.g. cromolyn or nedocromil) within the past 7 days
  * Other antihistamines or cough and cold preparations (with the exception of single ingredient guaifenesin products), or over-the-counter (OTC) sleep aid medications within the past 7 days
  * Systemic antibiotics within the past 7 days
  * Other concomitant medications that will interfere with the study, in the opinion of the investigator
* Previous participation in another clinical/pharmacological trial within the past month prior to V1
* Have already participated in this study or participated in this study at another site
* Children of any member of the study site staff
* Sibling with sleep apnea or sudden infant death syndrome (SIDS)
* Exposure to other conditions known to be potential risk factors for SIDS, such as but not limited to (this should be determined on a case by case basis taking into account the subject's entire medical history and environmental living conditions):

  * Mothers who smoked or abused drugs during pregnancy
  * Extremely young mothers (defined as age 19 or younger when pregnant)
  * Children currently exposed to a caregiver which is a heavy cigarette smoker (defined as smoking at least a pack of cigarettes per day)
  * Babies who sleep regularly on their face or are not put to sleep on their backs
  * Premature birth gestational age ≤ 37 weeks) or low birth weight (below 10 percentile for gestational age)

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (26):
- United States (26):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Crescent City, California
  - Huntington Beach, California
  - Los Angeles, California
  - Orange, California
  - Roseville, California
  - Stockton, California
  - Albany, Georgia
  - Gainesville, Georgia
  - Normal, Illinois
  - Bridgeton, Missouri
  - Omaha, Nebraska
  - Oklahoma City, Oklahoma
  - Barnwell, South Carolina
  - Spartanburg, South Carolina
  - Kingsport, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - San Antonio, Texas
  - Sugarland, Texas
  - Richmond, Virginia

REFERENCES:
- [Derived] Hampel F, Ratner P, Haeusler JM. Safety and tolerability of levocetirizine dihydrochloride in infants and children with allergic rhinitis or chronic urticaria. Allergy Asthma Proc. 2010 Jul-Aug;31(4):290-5. doi: 10.2500/aap.2010.31.3349. PMID 20819318
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was randomized to levocetirizine but received placebo; hence the number of subjects in both treatment groups in the Safety Population differs by 1 from the number of the subjects randomized (STARTED) to the respective treatment group. All results are presented for the safety population for which the subjects were analyzed as treated.
Groups:
- Placebo: Placebo (5 drops) dosed by mouth in the morning at breakfast time once a day for 2 weeks from Visit 2 (Day 0) to Visit 4 (Day 14) or the Early Discontinuation Visit (EDV).
- Levocetirizine: Levocetirizine dihydrochloride 1.25 mg oral drops (5 drops containing 5 mg/mL) dosed by mouth in the morning at breakfast time once a day for 2 weeks from Visit 2 (Day 0) to Visit 4 (Day 14) or the Early Discontinuation Visit (EDV).
Period: Overall Study
Arm/Group | Placebo | Levocetirizine
Started | 23 | 46 (One subject was randomized to levocetirizine but received placebo.)
Safety Population | 24 | 45 (Subjects in the Safety Population were analyzed as treated.)
Completed | 22 | 43
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Levocetirizine | Total
Number analyzed (Participants) | 24 | 45 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 45 | 69
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.03 (1.80) | 8.87 (1.63) | 8.93 (1.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 11 | 28 | 39
Region of Enrollment [Number; unit: participants]
  United States | 24 | 45 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Ventricular Rate (VR)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 20 | 38
beats per minute | -7.6 (17.3) | -4.0 (16.9)

2. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in RR Interval
Description: The RR interval refers to the respective time interval in the Electrocardiogram (ECG)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 20 | 38
milliseconds | 28.0 (63.9) | 14.9 (58.4)

3. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in PR Interval
Description: The PR interval refers to the respective time interval in the Electrocardiogram (ECG)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 20 | 38
milliseconds | 0.8 (11.3) | 3.1 (11.3)

4. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in QRS Duration
Description: The QRS duration refers to the respective time interval in the Electrocardiogram (ECG)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 20 | 38
milliseconds | 1.4 (6.4) | 0.3 (5.7)

5. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in QT Interval
Description: The QT interval refers to the respective time in the Electrocardiogram (ECG)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 20 | 38
milliseconds | 4.5 (21.1) | -0.3 (18.7)

6. Primary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF)
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 20 | 38
milliseconds | -1.3 (20.9) | -3.9 (17.3)

7. Primary Outcome: Absolute Value of QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) at Visit 3 (Day 7)
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG)
Time Frame: 7 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 21 | 42
milliseconds | 360.3 (15.2) | 354.5 (21.1)

8. Primary Outcome: Absolute Value of QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF) at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV)
Description: The QT interval refers to the respective time interval in the Electrocardiogram (ECG)
Time Frame: 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 23 | 39
milliseconds | 355.3 (17.7) | 351.9 (18.0)

9. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Total Bilirubin
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: micromole per liter [µmol/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 19 | 35
micromole per liter [µmol/L] | 0.000 [-1.71 to 1.71] | 0.000 [-3.42 to 3.42]

10. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Alanine Aminotransferase (ALT)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: unit per liter [U/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 19 | 34
unit per liter [U/L] | -2.0 [-27 to 15] | -1.0 [-24 to 41]

11. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Aspartate Aminontransferase (AST)
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: unit per liter [U/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 19 | 34
unit per liter [U/L] | 2.0 [-15 to 21] | -1.0 [-36 to 23]

12. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Blood Urea Nitrogen
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: millimole per liter [mmol/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 19 | 36
millimole per liter [mmol/L] | 0.0000 [-0.714 to 2.856] | 0.0000 [-3.927 to 4.641]

13. Secondary Outcome: Change From Baseline at Visit 4 (Day 14) or at Early Discontinuation Visit (EDV) in Blood Creatinine
Time Frame: Baseline, 14 days
Population: Safety Population; only non-missing values were analyzed
Measure: Median (Full Range); unit: micromole per liter [μmol/L]
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 19 | 36
micromole per liter [μmol/L] | -0.8840 [-9.724 to 20.332] | -0.8840 [-18.564 to 10.608]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Visit 1 (Day -2 to -28) over randomization and On-treatment Period up to the Follow-up Visit (Day 21±2).
Description: Adverse Events refer to the Safety Population including all subjects who were dispensed study medication at least once.
Arm/Group | Placebo | Levocetirizine
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/45
Other Adverse Events (participants affected / at risk) | 17/24 | 29/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Levocetirizine (N=45)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | Levocetirizine (N=45)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (6)
Teething (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 7 (7)
Irritability (General disorders) | 3 (3) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Heat rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.